CLINICAL TRIAL: NCT06465186
Title: Phase 2a Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Efinopegdutide (MK-6024) in Adults With Compensated Cirrhosis Secondary to Metabolic Dysfunction-Associated Steatohepatitis
Brief Title: A Clinical Study of Efinopegdutide in People With Compensated Cirrhosis Due to Steatohepatitis (MK-6024-017)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6024-017; 2024-510923-20-00 (Registry Identifier: EU CT); MK-6024-017 (Other: MSD); jRCT2031240217 (Registry Identifier: jRCT); U1111-1302-7589 (Registry Identifier: UTN)
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Non-alcoholic Fatty Liver Disease; Nonalcoholic Steatohepatitis; NAFLD; Metabolic Dysfunction-associated Steatotic Liver Disease; Metabolic Dysfunction-associated Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Efinopegdutide (Experimental): Participants will start efinopegdutide once a week at the lowest dose level. Then, the dose level will go up every month for three months until they are getting the highest dose level. Efinopegdutide is given as an injection under the skin (subcutaneous injection) for 28 weeks.
  Interventions: Combination Product: Efinopegdutide
- Placebo (Placebo Comparator): Participants will receive placebo once a week. A placebo looks like the study medicine but has no study medicine in it. Using a placebo helps researchers better understand the effects of a study medicine.
  Placebo is given as an injection under the skin (subcutaneous injection) for 28 weeks.
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Combination Product: Efinopegdutide — Efinopegdutide is given as a subcutaneous injection using a single-use prefilled syringe, once per week for 28 weeks
  Other Names: MK-6024
  Arms: Efinopegdutide
Combination Product: Placebo — Placebo is given as a subcutaneous injection using a single-use prefilled syringe once per week for 28 weeks.
  Arms: Placebo

SUMMARY:
Researchers are looking for ways to treat a type of liver disease caused by elevated liver fat, called metabolic dysfunction-associated steatohepatitis (MASH). MASH was formerly called non-alcoholic steatohepatitis (NASH). Researchers want to learn if a study medicine called efinopegdutide can treat MASH.The goals of this study are to learn:

* If efinopegdutide can lower the amount of fat, inflammation, and scarring (fibrosis) in the liver
* About the safety of efinopegdutide and how well people tolerate it

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has compensated cirrhosis caused by metabolic dysfunction-associated steatohepatitis (MASH)
* Has either type 2 diabetes that is controlled by diet or medication, or does not have type 2 diabetes

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has history of a liver disease other than MASH, for example, Hepatitis B or C, drug-induced liver disease, or autoimmune liver disease
* Has history of type 1 diabetes
* Had a bariatric surgical procedure less than 5 years before entry into the study
* History of pancreatitis
* Major illnesses like recent (within 6 months of study entry) episodes of heart problems, such as congestive heart failure, unstable angina, heart attack, stroke, or mini-stroke

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2026-08-06 (Estimated); Study Completion 2026-08-06 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Liver Fat Content (LFC) at Week 28 | Baseline and 28 weeks
  Researchers will measure the change in the amount of fat in the liver using magnetic resonance imaging (MRI) after about 7 months of treatment.
  The change in MRI-Estimated proton density fat fraction (PDFF) will be measured from baseline to 28 weeks.
Percentage of Participants Who Experienced an Adverse Event (AE) | Up to approximately 36 weeks
  An AE is a health problem that happens or worsens during the study
Percentage of Participants Discontinuing Study Medication Due to an AE | Up to approximately 28 weeks
  An AE is a health problem that happens or worsens during a study. The percentage of participants who stop study treatment due to an AE will be reported.

SECONDARY OUTCOMES:
Change from Baseline in Iron-corrected T1 (cT1) at Week 28 | Baseline and up to 28 Weeks
  Researchers will measure the change in liver inflammation and scarring (fibrosis) after about 7 months of treatment.
  MRI measurement of cT1 mapping will be used to indicate the amount of liver inflammation and fibrosis. The change in cT1 mapping from baseline to 28 weeks will be presented.
Change from Baseline in Enhanced Liver Fibrosis (ELF) score at Week 28 | Baseline and up to 28 weeks
  Researchers will measure the change in liver scarring using biomarkers. Biomarkers are substances measured in blood that show normal or abnormal activity taking place in the liver.
  ELF is calculated using 3 markers of hepatic extracellular matrix turnover to generate a unitless numerical score. The change from baseline in ELF up to 28 weeks will be reported.
Change from Baseline in Propeptide of Type III Collagen (Pro-C3) at Week 28 | Baseline and up to 28 weeks
  Researchers will measure the change in liver scarring using biomarkers.
  Pro-C3 is measured in serum; Increasing levels indicate worsening of fibrosis activity. The change in Pro-C3 from baseline to 28 weeks will be reported.
Change from Baseline in Fibrosis-4 index (FIB-4) at Week 28 | Baseline and up to 28 weeks
  Researchers will measure the change in liver scarring using biomarkers.
  FIB-4 index is calculated using the participant's age and 3 serum markers (alanine aminotransferase [ALT], aspartate aminotransferase [AST], and platelet count). The change from baseline in FIB-4 after 28 weeks will be reported.
Change from Baseline in Liver Stiffness Measurement (LSM) Assessed by Vibration-controlled Transient Elastography (VCTE) at week 28 | Baseline and up to 28 weeks
  Researchers will measure the change in liver scarring using ultrasound.
  LSM is measured using VCTE. The change from baseline in LSM after 28 weeks will be reported.
Percent Change from Baseline in Body Weight at Week 28 | Baseline and up to approximately 28 weeks
  Body weight will be measured using a standardized, digital scale. The percent change from baseline in body weight after 28 weeks will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (68):
- United States (33):
  - The Institute for Liver Health II dba Arizona Clinical Trial-The Institute for Liver Health ( Site 0149), Chandler, Arizona
  - Arizona Clinical Trials ( Site 0158), Flagstaff, Arizona
  - The Institute for Liver Health II dba Arizona Liver Health - Peoria ( Site 0120), Peoria, Arizona
  - The Institute for Liver Health II dba Arizona Liver Health-Tucson ( Site 0111), Tucson, Arizona
  - California Liver Research Institute ( Site 0113), Pasadena, California
  - Acclaim Clinical Research ( Site 0137), San Diego, California
  - Velocity Clinical Research, Panorama City ( Site 0124), Van Nuys, California
  - Rocky Mountain Gastroenterology ( Site 0127), Littleton, Colorado
  - Synergy Healthcare ( Site 0118), Bradenton, Florida
  - Homestead Associates in Research, Inc. ( Site 0139), Homestead, Florida
  - Florida Research Institute ( Site 0116), Lakewood Rch, Florida
  - Floridian Clinical Research, LLC ( Site 0109), Miami Lakes, Florida
  - Southeast Clinical Research Center ( Site 0119), Dalton, Georgia
  - Delta Research Partners ( Site 0160), Bastrop, Louisiana
  - Louisiana Research Center ( Site 0161), Shreveport, Louisiana
  - Woodholme Gastroenterology Associates-Woodholme Gastroenterology Associates ( Site 0130), Glen Burnie, Maryland
  - Velocity Clinical Research Rockville ( Site 0143), Rockville, Maryland
  - Huron Gastroenterology ( Site 0102), Ypsilanti, Michigan
  - The Machuca Foundation ( Site 0115), Las Vegas, Nevada
  - Excel Clinical Research, LLC ( Site 0101), Las Vegas, Nevada
  - Southwest Gastroenterology Associates ( Site 0129), Albuquerque, New Mexico
  - Coastal Research Institute - Fayetteville ( Site 0159), Fayetteville, North Carolina
  - Lucas Research, Inc ( Site 0105), Morehead City, North Carolina
  - Texas Clinical Research Institute ( Site 0126), Arlington, Texas
  - Pinnacle Clinical Research ( Site 0104), Austin, Texas
  - Pinnacle Clinical Research-Corpus Christi ( Site 0156), Corpus Christi, Texas
  - Zenos Clinical Research ( Site 0136), Dallas, Texas
  - GI Alliance Department of Research ( Site 0162), Fort Worth, Texas
  - Houston Research Institute ( Site 0172), Houston, Texas
  - Houston Research Institute ( Site 0117), Houston, Texas
  - American Research Corporation ( Site 0131), San Antonio, Texas
  - Pinnacle Clinical Research-Clinical Research Coordination ( Site 0125), San Antonio, Texas
  - University of Virginia Health System ( Site 0164), Charlottesville, Virginia
- Australia (2):
  - Flinders Medical Centre-Hepatology and Liver Transplant Medicine ( Site 1202), Adelaide, South Australia
  - St Vincent's Hospital-Gastroenterology Department ( Site 1205), Melbourne, Victoria
- Canada (2):
  - Toronto General Hospital ( Site 0207), Toronto, Ontario
  - Diex Recherche Quebec ( Site 0204), Québec, Quebec
- Colombia (2):
  - Fundacion Santa Fe de Bogota ( Site 0403), Bogotá, Cundinamarca
  - Fundación Valle del Lili ( Site 0402), Cali, Valle del Cauca Department
- France (5):
  - Centre Hospitalier Universitaire de Nice - Hôpital l'Archet-Pôle de Référence Hépato Gastro-entérol ( Site 0704), Nice, Alpes-Maritimes
  - CHU Bordeaux Haut-Leveque-Service d'Hépato-gastroentérologie ( Site 0701), Pessac, Aquitaine
  - Hôpital de la Croix Rousse-Centre de Recherche Clinique ( Site 0705), Lyon, Auvergne-Rhône-Alpes
  - Hôpital Beaujon-Hépatologie ( Site 0703), Clichy, Hauts-de-Seine
  - Centre Hospitalier Universitaire de Limoges - Hôpital Dupuytren-Hépato-gastroentérologie ( Site 0702), Limoges, Limousin
- Israel (5):
  - Rambam Health Care Campus ( Site 0801), Haifa
  - Carmel Hospital-Liver Unit ( Site 0802), Haifa
  - Shaare Zedek Medical Center ( Site 0805), Jerusalem
  - Maccabi Health Services - Petah Tikva ( Site 0804), Petah Tikva
  - Assuta Medical Center ( Site 0806), Tel Aviv
- Japan (5):
  - Shinyurigaoka General Hospital ( Site 1401), Kawasaki, Kanagawa
  - Yokohama City University Hospital ( Site 1402), Yokohama, Kanagawa
  - University Hospital,Kyoto Prefectural University of Medicine ( Site 1404), Kyoto
  - Osaka Metropolitan University Hospital ( Site 1403), Osaka
  - Saga University Hospital ( Site 1405), Saga
- Puerto Rico (2):
  - ISIS CLINICAL RESEARCH CENTER ( Site 0606), Guaynabo
  - Klinical Investigations Group-Clinical Research ( Site 0601), San Juan
- Spain (8):
  - Hospital Universitario Marqués de Valdecilla-Gastroenterology and Hepatology ( Site 1004), Santander, Cantabria
  - Hospital Clínico Universitario de Valladolid-Servicio de Endocrinologia y Nutricion ( Site 1008), Valladolid, Castille and León
  - Hospital General de Tomelloso-Aparato Digestivo ( Site 1006), Tomelloso, Ciudad Real
  - CHUAC-Complejo Hospitalario Universitario A Coruña-Endocrinología ( Site 1007), A Coruña, La Coruna
  - CHUS - Hospital Clinico Universitario ( Site 1011), Santiago de Compostela, La Coruna
  - Hospital Universitari Vall d'Hebron-Liver Unit - Department of Internal Medicine ( Site 1002), Barcelona
  - Hospital Universitario La Paz-HEPATOLOGIA ( Site 1005), Madrid
  - HOSPITAL UNIVERSITARIO VIRGEN DEL ROCIO-Unidad de Ensayos clinicos de Aparato Digestivo ( Site 1001), Seville
- Thailand (2):
  - Chulalongkorn University ( Site 1301), Bangkok, Bangkok
  - Faculty of Medicine Siriraj Hospital-Department of Medicine ( Site 1302), Bangkok, Bangkok
- United Kingdom (2):
  - King's College Hospital ( Site 1104), London, London, City of
  - Aberdeen Royal Infirmary-Department of Gastroenterology ( Site 1102), Aberdeen, Scotland

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26278&tenant=MT_MSD_9011